CLINICAL TRIAL: NCT00000981
Title: Efficacy and Safety of Oral FIAC in AIDS Patients With Cytomegalovirus Infection: A Dose Ranging Study
Brief Title: The Safety and Effectiveness of FIAC in the Treatment of Cytomegalovirus (CMV) in Patients With AIDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Oclassen Pharmaceuticals (Industry)
Purpose: Treatment
Other Study IDs: ACTG 122 FIAC; R89-001-01, 02, 03, 04
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Cytomegalovirus Infections; HIV Infections
Keywords: Retinitis; AIDS-Related Opportunistic Infections; Pyrimidine Nucleosides; Drug Evaluation; fiacitabine; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome; Antiviral Agents
MeSH Terms: conditions — Cytomegalovirus Infections; HIV Infections; Retinitis; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — fiacitabine

INTERVENTIONS:
Drug: Fiacitabine

SUMMARY:
To find oral doses of FIAC (a pyrimidine nucleoside analog) that are effective in treating cytomegalovirus (CMV) viremia in HIV-infected immunocompromised patients; to determine tolerance and safety of FIAC in this patient population; and to determine pharmacokinetics following multiple doses of FIAC. (An example of another nucleoside analog effective against retroviruses such as HIV is zidovudine (AZT).) CMV infection is a medically significant opportunistic disease in patients with HIV-related infection. The purine nucleoside ganciclovir has been used to treat AIDS patients with CMV disease. Although ganciclovir is useful in treating CMV disease, such treatment is frequently complicated by hematologic (blood) toxicity. Also, treatment is difficult because it requires daily intravenous dosing. Test tube studies show that FIAC and its primary breakdown product FIAU are highly and specifically active against several viruses including CMV. A single-dose, pharmacokinetic (blood level) study showed that FIAC, when taken orally, is readily absorbed into the bloodstream, and most of it is converted to FIAU.

DETAILED DESCRIPTION:
CMV infection is a medically significant opportunistic disease in patients with HIV-related infection. The purine nucleoside ganciclovir has been used to treat AIDS patients with CMV disease. Although ganciclovir is useful in treating CMV disease, such treatment is frequently complicated by hematologic (blood) toxicity. Also, treatment is difficult because it requires daily intravenous dosing. Test tube studies show that FIAC and its primary breakdown product FIAU are highly and specifically active against several viruses including CMV. A single-dose, pharmacokinetic (blood level) study showed that FIAC, when taken orally, is readily absorbed into the bloodstream, and most of it is converted to FIAU.

Patients are treated as outpatients if general health permits. This is continued for up to 90 days or until failure on basis of efficacy, tolerance, or toxicity. The dose escalation between groups of patients uses the formula n + 0.7n. Entry of new patients at the next higher dose is based on results of antiviral, tolerance, and safety data for the prior cohort when they have received at least 14 days of therapy. Consecutively qualifying patients are enrolled for each dose group and not based on either disease severity or expected tolerance. Although not formally randomized due to the sequential nature of the study and serious medical condition of the patients, every attempt to avoid bias in assigning a patient to a dose is made. Patients are advised to avoid heavy exercise within 24 hours of any laboratory tests.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Pentamidine aerosol for prophylaxis of recurrent Pneumocystis carinii pneumonia (PCP) in patients currently receiving such treatment.

Prior Medication:

Allowed:

* Zidovudine (AZT) but only if patient has been taking the drug for > 6 weeks at a dose = or < 600 mg/day, and had < 10 percent decrease in hematocrit, neutrophils, and platelets in the last 30 days. Those off AZT must have been off it for > 1 month.

Patients must:

* Have documented cytomegalovirus (CMV) viremia or viruria.
* Have a diagnosis of HIV infection by ELISA or Western blot.
* Be able to participate as an outpatient.
* Be ambulatory.
* Grade 0 or 1 AIDS Clinical Trial Group toxicity grades for specified laboratory tests.
* Be competent to sign informed consent.
* Be able to cooperate with the treatment plan and evaluation schedule.

NOTE:

* The screening tests must be initiated and completed within 4 weeks prior to the first dose of FIAC.

Concomitant diseases allowed:

* Stable mucocutaneous Kaposi's sarcoma.
* Superficial or uncomplicated infections such as thrush.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* HIV wasting syndrome (involuntary weight loss > 10 percent of baseline body weight and/or chronic diarrhea or weakness and documented fever for at least 30 days).
* Clinical or x-ray evidence of bronchitis, pneumonitis, pulmonary edema, effusion, or suspected active tuberculosis.
* Any unstable medical condition including serious cardiovascular, infectious, oncologic, renal, or hepatic condition.
* Cytomegalovirus end organ disease.
* Kaposi's sarcoma requiring chemotherapy.
* Systemic fungal infection requiring amphotericin therapy.
* Diagnosis of idiopathic thrombocytopenic purpura (persistent platelet counts < 100000 platelets/mm3 for = or > 3 months).

Patients with the following are excluded:

* HIV wasting syndrome.
* Clinical or x-ray evidence of bronchitis, pneumonitis, pulmonary edema, effusion, or suspected active tuberculosis.
* Any unstable medical condition including serious cardiovascular, infectious, oncologic, renal, or hepatic condition.
* Cytomegalovirus (CMV) end organ disease e.g., retinitis, hepatitis, gastroenteritis.

Prior Medication:

Excluded within 4 weeks of study entry:

* Zidovudine (AZT).
* Acyclovir.
* Ganciclovir (DHPG).
* Foscarnet.
* Interferon.
* Other drug with putative anticytomegaloviral activity.
* Any immunostimulating drug not specifically allowed.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78
Dates: Study Completion 1993-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Natl Institute of Health, Bethesda, Maryland
  - Univ of Washington / Madison Clinic, Seattle, Washington